CLINICAL TRIAL: NCT01894334
Title: Mechanism and Early Intervention Research on Acute Lung Injury During Emergence Surgery of Acute Stanford A Aortic Dissection
Brief Title: Mechanism and Early Intervention Research on ALI During Emergence Surgery of Acute Stanford A Aortic Dissection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Principal Investigator, WeiPing Cheng, Professor；Chief Physician, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2011-2006-03
Record Dates: First submitted 2013-06-08; First posted 2013-07-10 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Acute Aortic Dissection
Keywords: Aortic dissection; acute lung injury; injury mechanism; early intervention
MeSH Terms: conditions — Aortic Dissection; Acute Lung Injury | interventions — urinastatin; Tranexamic Acid; Edaravone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control group (No Intervention): no intervention
- Tranexamic acid group (Experimental): tranexamic acid ，intravenous 30mg/kg/d，Preoperative
  Interventions: Drug: Tranexamic acid
- Edaravone group (Experimental): edaravone, iv, 1mg/kg/d,Preoperative
  Interventions: Drug: Edaravone
- Ulinastatin group (Experimental): Ulinastatin ,iv，20,000 U /kg/d，Preoperative
  Interventions: Drug: Ulinastatin

INTERVENTIONS:
Drug: Ulinastatin
  Arms: Ulinastatin group
Drug: Tranexamic acid
  Arms: Tranexamic acid group
Drug: Edaravone
  Arms: Edaravone group

SUMMARY:
The morbidity rate of Stanford A type Acute Aortic Dissection（AAD） has been increasing, about 5-10/100,000* per year. Emergency surgery has been the main treatment for Acute Aortic Dissection, however perioperative mortality rate can be as high as 15~30%. Acute lung injury (ALI) is one of the main complications that happen during the perioperative period, which by itself covers 30%-50% of the overall mortality rate. Both domestic and foreign countries lack researches on risk factors, pathogenesis, disease progression and outcome of ALI, which happen during the perioperative period of Acute Aortic Dissection patients.

This topic study follow projects in the preoperative of Acute Aortic Dissection'surgery

1. hemodynamic changes (aortic dissection resulting in acute aortic regurgitation, cardiac tamponade and proximal high blood pressure)
2. ischemia - reperfusion injury of aortic dissection distal organ
3. Aortic intima-media exposure cause coagulation / fibrinolytic system function disorder
4. systemic inflammatory response syndrome; use relevant clinical radiographic parameters, indicators of respiratory mechanics (oxygenation index and lung injury index) and biochemical indicators.

To discuss risk factors and possible mechanisms of ADD patients with pre-operative ALI and observe their influences on the progress and prognosis of AAD, to explore early intervention in the preoperative for possible risk factors and mechanisms and to evaluate their influences on the prognosis, to achieve the purpose of reducing AAD perioperative mortality of ALI and medical expenses.

ELIGIBILITY:
Inclusion Criteria:

* AAD patients within 48 hrs of onset who are prepared for aortic surgery
* Age between 18 and 70
* Willing to sign the informed consent

Exclusion Criteria:

* A history of chronic respiratory disease before onset
* A history of chronic heart failure or coronary heart disease before onset
* A history of chronic liver or kidney dysfunction before onset
* Severe central nervous system syndrome after admission
* Refuse to sign the informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
perioperative outcome and improve of ALI | Period from 48 hours before surgery to 12 hours after ICU
  indicators
  * chest imaging (preoperative, 12 hours after ICU);
  * arterial blood gases and alveolar-arterial oxygen difference (before surgery, and immediately after induction of anesthesia, before surgery ends and 12 hours after ICU);
  * respiratory mechanics (immediately after induction of anesthesia, before the end of surgery and 12 hours after ICU); including peak airway pressure, plateau pressure, dynamic and static compliance and so on.

SECONDARY OUTCOMES:
systemic inflammatory response | Period from 48 hours before surgery to 12 hours after ICU
  Indicators
  * Lung lavage (immediately after induction of anesthesia、before the end of surgery)
  * determination of imflammatory cytokines (IL-6, IL-8, Tumor Necrosis Factor -α, Cluster of Differentiation 11 /Cluster of Differentiation 18 , myeloperoxidase) and surface-active substance

CONTACTS AND LOCATIONS:
Overall Officials: WeiPing Cheng, master, Principal Investigator — Chief Physician，Professor

REFERENCES:
- [Derived] Gao Z, Pei X, He C, Wang Y, Lu J, Jin M, Cheng W. Oxygenation impairment in patients with acute aortic dissection is associated with disorders of coagulation and fibrinolysis: a prospective observational study. J Thorac Dis. 2019 Apr;11(4):1190-1201. doi: 10.21037/jtd.2019.04.32. PMID 31179061
- [Derived] Pan X, Lu J, Cheng W, Yang Y, Zhu J, Jin M. Independent factors related to preoperative acute lung injury in 130 adults undergoing Stanford type-A acute aortic dissection surgery: a single-center cross-sectional clinical study. J Thorac Dis. 2018 Jul;10(7):4413-4423. doi: 10.21037/jtd.2018.06.140. PMID 30174890
- [Derived] Cheng Y, Jin M, Dong X, Sun L, Liu J, Wang R, Yang Y, Lin P, Hou S, Ma Y, Wang Y, Pan X, Lu J, Cheng W. Mechanism and early intervention research on ALI during emergence surgery of Stanford type-A AAD: Study protocol for a prospective, double-blind, clinical trial. Medicine (Baltimore). 2016 Oct;95(42):e5164. doi: 10.1097/MD.0000000000005164. PMID 27759648